CLINICAL TRIAL: NCT03865433
Title: The Effect of a Sub-symptom Threshold Aerobic Exercise Program on Recovery in Concussed Athletes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rocky Mountain University of Health Professions (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Emily Kosderka, Principle Investigator, Rocky Mountain University of Health Professions
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ConcussionRecovery2019
Record Dates: First submitted 2019-02-27; First posted 2019-03-06 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Concussion, Mild; Rehabilitation
MeSH Terms: conditions — Brain Concussion | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to one of two groups: the intervention group or the placebo/control group
Who Masked: Care Provider
Masking Description: Study physicians will be blinded to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): Intervention: aerobic exercise Subjects in the exercise group will be prescribed exercise at a target heart rate (THR) of approximately 80% of the achieved heart rate during the Buffalo Concussion Treadmill Test (BCTT). They will be given this prescription in writing to provide to their athletic trainer. Subjects will complete 30 minutes of daily exercise (including 5 minutes of warm up and 5 minutes of cool down) on an exercise bike or walking and supervised by an athletic trainer. This program may be modified by increasing heart rate threshold 5-10 beats per minute per week by the athletic trainer as the heart rate for symptom exacerbation increases.
  Interventions: Other: Aerobic Exercise
- Placebo/Stretching (Placebo Comparator): Intrvention: stretching program Subjects assigned to the Stretching/Placebo group will be given a stretching protocol and instructions to report to their athletic trainer on a daily basis as soon as possible. . Subjects will then complete a 15-25 minute stretching program under supervision by the athletic trainer or other designated research personnel. The stretching protocol will be progressive and will change weekly as subjects continue their recovery.
  Interventions: Other: Placebo/Stretching

INTERVENTIONS:
Other: Aerobic Exercise — Sub-symptom threshold aerobic exercise at a dose of 30 minutes per day, five days per week.
  Arms: Exercise Group
Other: Placebo/Stretching — A detailed, progressive stretching program to be performed for approximately 20-30 minutes per day, five days per week
  Arms: Placebo/Stretching

SUMMARY:
The purpose of this randomized controlled trial is to examine whether systematic sub-threshold exercise is effective in improving recovery time in athletes after sport related concussion (SRC) compared to those who participate in a placebo/stretching protocol. subjects will be randomized into either an Exercise group or a Placebo/stretching group. subjects in the Exercise group will participate in an individualized exercise program supervised by their athletic trainer while the Placebo/stretching group will engage in a standardized stretching routine supervised by their athletic trainer throughout the duration of their recovery.

Hypothesis 1: subjects in the aerobic Exercise group will require fewer days to recover from SRC than those who follow a placebo/stretching protocol.

Hypothesis 2: heart rate threshold (HRt) achieved on the graded treadmill test will be associated with days to recovery (i.e., the lower the HRt, the longer the time to recovery).

Hypothesis 3: Vestibular Ocular Motor Screen (VOMS) performance will be indicative of time to clinical recovery from concussion as evidenced by a strong correlation between VOMS score and days to clinical recovery.

Hypothesis 4: Sub-threshold aerobic exercise will facilitate improvement in VOMS post-concussion.

Hypothesis 5: subjects in the aerobic exercise group will demonstrate greater dynamic stability as evidenced by greater reach in each of the 3 primary directions (anterior, posterior medial and posterior lateral) for their right and left lower extremity.

DETAILED DESCRIPTION:
For this randomized controlled trial, a random number generator will be used to randomly assign subjects to either the Placebo/Stretching group or the Exercise group. Study physicians will be blinded to group assignment. Each subject will be given a subject ID number and will complete a brief medical history. They will then be escorted by a designated health care professional who is either the site-coordinator or another health care provider trained in the administration of the Buffalo Concussion Treadmill Test (BCTT) to the treadmill. There, they will be fitted with an ActiGraph activity monitor to be worn throughout their recovery period. The ActiGraph is a small, non-invasive unit that measures human rest and activity cycles. It will be worn similarly to a wrist watch and secured in place with a disposable wristband. Resting heart rate variability (HRV) will be assessed using the Elite HRV app for smartphone. Trained research personnel will assist the subject with fitting the Polar H7 heart rate sensor and finding a comfortable seated position. The heart rate sensor will then connect with the Elite HRV app for smart phone. Once connected, it will take approximately 2 minutes to record the data. Subjects will complete the BCTT in the clinic at the first available testing session no earlier than 48 hours following injury. VOMS and Y-Balance test will also be administered and recorded.

Stretching/Placebo Group Subjects assigned to the Stretching/Placebo group will be given a stretching protocol and instructions to report to their athletic trainer on a daily basis as soon as possible. Prior to the beginning of each intervention session, subjects will be assessed using standard of care protocols which include verbal feedback, symptom scale, and visual-analog scale (VAS). Subjects with a self-reported VAS of ≥7 will not stretch that day. Subjects with a score of ≤ 6 will then complete a 15-25 minute stretching program under supervision by the athletic trainer or other designated research personnel. Following completion of the stretching program for that day, the athletic trainer will record exercise duration and heart rate (HR) (as monitored by the Polar H7 Heart Rate Sensor). The stretching protocol will be progressive and will change weekly as subjects continue their recovery.

Exercise Group Subjects in the exercise group will be prescribed exercise at a target heart rate (THR) of approximately 80% of the achieved heart rate during the BCTT. They will be given this prescription in writing to provide to their athletic trainer. Prior to the beginning of each intervention session, subjects will be assessed using standard of care protocols which include verbal feedback, symptom scale, and visual-analog scale. Subjects with a self-reported Visual Analog Scale (VAS) of ≥ 7 will not exercise that day. Subjects with a score of ≤ 6 will then complete 30 minutes of daily exercise (including 5 minutes of warm up and 5 minutes of cool down) on an exercise bike or walking and supervised by an athletic trainer. Subjects will be instructed to terminate exercise at the first sign of symptom exacerbation or after 30 minutes, whichever occurs first. Athletic trainers will instruct subjects to cease exercise if additional symptoms appear or if symptoms worsen. This program may be modified by increasing heart rate threshold 5-10 beats per minute per week by the athletic trainer as the heart rate for symptom exacerbation increases. The supervising athletic trainer will record exercise duration and THR (as monitored by the Polar H7 Heart Rate Sensor).

Due to medical ethics, subjects will undergo any other individualized rehabilitation recommendations made by the physician or treating physical therapist throughout their individual treatment period. Common rehabilitation interventions include vestibular, oculomotor, cervicogenic, and balance exercises. Subjects may undergo one or all of these depending on their individual needs. Therefore, the exercise protocol identified in this application is a supplement to their standard care provided by medical personnel.

All Subjects All subjects will complete the Symptom Form daily for the duration of their symptom presentation. In addition to reporting to their athletic trainer, subjects will be provided with a link to a secured website on which they will be asked to enter their symptoms at approximately the same time each evening. An option will be to provide the surveys and envelopes to complete these in hard copy.

When symptoms are no longer reported to the athletic trainer by the subject, the athletic trainer will complete the clinical battery associated with their respective concussion protocol prior to the subject's appointment with the study physician to seek clearance for return to play. The study physician will conduct a standardized physical exam and determine if the subject has met the following criteria for clinical recovery:

1. normal or baseline Standardized Assessment of Concussion;
2. normal neurological exam; and
3. can complete the BCTT without symptom exacerbation.
4. VOMS and Y-Balance

Prior to the clearance BCTT, subjects will have Heart Rate Variability (HRV) measured using the Elite HRV app for smart phone. Trained research personnel will assist the subject with fitting the Polar H7 heart rate sensor and finding a comfortable seated position. The heart rate sensor will then connect with the Elite HRV app for smartphone. Once connected, it will take approximately 2 minutes to record the data.

The subject will then begin at Stage 3 of the stepwise return to sport (RTS) strategy as outlined in the Berlin guidelines and full RTS will be allowed when the subject has completed each step of the stepwise RTS criteria without symptom exacerbation. Number of days from date of injury to full RTS (including days in the Berlin RTS) will be recorded, analyzed, and compared for the Placebo/Stretching group and the Exercise group.

ELIGIBILITY:
Inclusion Criteria:

1. are aged 13-17, years and a high school student-athlete who attends school where an athletic trainer can supervise the exercise protocol;
2. have sustained a concussion within 2-7 days of clinic presentation and diagnosed by a study physician;
3. demonstrate symptom exacerbation during a graded treadmill exercise test and cannot complete the test;
4. are currently participating in a school or club sport;
5. are English speaking and capable of giving assent

Exclusion Criteria:

1. have a reported history of neurological condition or disorder including but not limited to brain surgery, special education, seizure disorder, speech pathology, previous diagnosis of Post-Concussion Syndrome (PCS),
2. are unwilling to exercise,
3. have focal neurologic deficit that would represent risk for walking/running on treadmill,
4. exhibit an inability to exercise due to injury, known heart disease, or increased cardiac risk,
5. have experienced more than 3 previous concussions,
6. have suffered a substantial comorbidity (eg,cervical injury),
7. currently taking β-blockers, calcium channel blockers, or prophylactic headache medications (e.g., amitriptyline, topiramate), or
8. have a resting blood pressure of > 140/90.
9. If the potential participant or parent/guardian is unable to fully understand the study protocol or study risks due to injury or developmental delay, the potential participant will be excluded from the study.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Estimated)
Dates: Start 2019-02-27 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Time to full clinical recovery | 0-45 days
  days between injury and return to play

SECONDARY OUTCOMES:
Heart rate | Achieved HR measured and recorded on first Buffalo Concussion Treadmill Test (Week 0-baseline)-6 weeks
  Relationship between achieved heart rate on the Buffalo Concussion Test (Monitored using a Polar heart rate monitor) and recovery time.
Vestibular Ocular Motor Screening (VOMS) | Recorded on first visit (Week 0-baseline)-6 weeks
  Improved vestibular and oculo motor function with the treatment, as reflected by lower scores
Y Balance Test (YBT) score | Administered and recorded on the first visit (Week 0-baseline)-6 weeks
  Improved balance as indicated by increased reach scores with the treatment
Concussion symptom burden | Week 0 (baseline)- 6 weeks
  Improvement on The Post-Concussion Symptom Scale with the treatment, as indicated by lower scores

CONTACTS AND LOCATIONS:
Overall Officials: Emily Kosderka, MS, Principal Investigator — Rocky Mountain University of Health Professions; Douglas Powell, PhD, Study Chair — Rocky Mountain University of Health Professions
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McCrory P, Meeuwisse W, Dvorak J, Aubry M, Bailes J, Broglio S, Cantu RC, Cassidy D, Echemendia RJ, Castellani RJ, Davis GA, Ellenbogen R, Emery C, Engebretsen L, Feddermann-Demont N, Giza CC, Guskiewicz KM, Herring S, Iverson GL, Johnston KM, Kissick J, Kutcher J, Leddy JJ, Maddocks D, Makdissi M, Manley GT, McCrea M, Meehan WP, Nagahiro S, Patricios J, Putukian M, Schneider KJ, Sills A, Tator CH, Turner M, Vos PE. Consensus statement on concussion in sport-the 5th international conference on concussion in sport held in Berlin, October 2016. Br J Sports Med. 2017 Jun;51(11):838-847. doi: 10.1136/bjsports-2017-097699. Epub 2017 Apr 26. No abstract available. PMID 28446457
- [Background] Leddy JJ, Kozlowski K, Donnelly JP, Pendergast DR, Epstein LH, Willer B. A preliminary study of subsymptom threshold exercise training for refractory post-concussion syndrome. Clin J Sport Med. 2010 Jan;20(1):21-7. doi: 10.1097/JSM.0b013e3181c6c22c. PMID 20051730
- [Background] Thomas DG, Apps JN, Hoffmann RG, McCrea M, Hammeke T. Benefits of strict rest after acute concussion: a randomized controlled trial. Pediatrics. 2015 Feb;135(2):213-23. doi: 10.1542/peds.2014-0966. Epub 2015 Jan 5. PMID 25560444
- [Background] Leddy JJ, Willer B. Use of graded exercise testing in concussion and return-to-activity management. Curr Sports Med Rep. 2013 Nov-Dec;12(6):370-6. doi: 10.1249/JSR.0000000000000008. PMID 24225521
- [Background] Kurowski BG, Hugentobler J, Quatman-Yates C, Taylor J, Gubanich PJ, Altaye M, Wade SL. Aerobic Exercise for Adolescents With Prolonged Symptoms After Mild Traumatic Brain Injury: An Exploratory Randomized Clinical Trial. J Head Trauma Rehabil. 2017 Mar/Apr;32(2):79-89. doi: 10.1097/HTR.0000000000000238. PMID 27120294
- [Background] Maerlender A, Rieman W, Lichtenstein J, Condiracci C. Programmed Physical Exertion in Recovery From Sports-Related Concussion: A Randomized Pilot Study. Dev Neuropsychol. 2015;40(5):273-8. doi: 10.1080/87565641.2015.1067706. Epub 2015 Jul 31. PMID 26230745
- [Background] Schneider KJ, Iverson GL, Emery CA, McCrory P, Herring SA, Meeuwisse WH. The effects of rest and treatment following sport-related concussion: a systematic review of the literature. Br J Sports Med. 2013 Apr;47(5):304-7. doi: 10.1136/bjsports-2013-092190. PMID 23479489
- [Background] Buckley TA, Munkasy BA, Clouse BP. Acute Cognitive and Physical Rest May Not Improve Concussion Recovery Time. J Head Trauma Rehabil. 2016 Jul-Aug;31(4):233-41. doi: 10.1097/HTR.0000000000000165. PMID 26394292
- [Background] Grool AM, Aglipay M, Momoli F, Meehan WP 3rd, Freedman SB, Yeates KO, Gravel J, Gagnon I, Boutis K, Meeuwisse W, Barrowman N, Ledoux AA, Osmond MH, Zemek R; Pediatric Emergency Research Canada (PERC) Concussion Team. Association Between Early Participation in Physical Activity Following Acute Concussion and Persistent Postconcussive Symptoms in Children and Adolescents. JAMA. 2016 Dec 20;316(23):2504-2514. doi: 10.1001/jama.2016.17396. PMID 27997652
- [Background] Polak P, Leddy JJ, Dwyer MG, Willer B, Zivadinov R. Diffusion tensor imaging alterations in patients with postconcussion syndrome undergoing exercise treatment: a pilot longitudinal study. J Head Trauma Rehabil. 2015 Mar-Apr;30(2):E32-42. doi: 10.1097/HTR.0000000000000037. PMID 24721808
- [Background] Baker JG, Freitas MS, Leddy JJ, Kozlowski KF, Willer BS. Return to full functioning after graded exercise assessment and progressive exercise treatment of postconcussion syndrome. Rehabil Res Pract. 2012;2012:705309. doi: 10.1155/2012/705309. Epub 2012 Jan 16. PMID 22292122
- [Background] Gagnon I, Galli C, Friedman D, Grilli L, Iverson GL. Active rehabilitation for children who are slow to recover following sport-related concussion. Brain Inj. 2009 Nov;23(12):956-64. doi: 10.3109/02699050903373477. PMID 19831492
- [Background] Cordingley D, Girardin R, Reimer K, Ritchie L, Leiter J, Russell K, Ellis MJ. Graded aerobic treadmill testing in pediatric sports-related concussion: safety, clinical use, and patient outcomes. J Neurosurg Pediatr. 2016 Dec;25(6):693-702. doi: 10.3171/2016.5.PEDS16139. Epub 2016 Sep 13. PMID 27620871